CLINICAL TRIAL: NCT03418571
Title: A Randomized, Double-blind, Multicenter, Multiple-dose Study of ALX-0171 Versus Placebo Along With Standard of Care in Japanese Infants and Young Children Hospitalized for Respiratory Syncytial Virus Lower Respiratory Tract Infection
Brief Title: Evaluation of ALX-0171 in Japanese Children Hospitalized for Respiratory Syncytial Virus Lower Respiratory Tract Infection
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: The Sponsor decided to discontinue ALX-0171 development (due to insufficient evidence of efficacy). As a result, the ALX0171-C203 study was early terminated.
Sponsor: Ablynx, a Sanofi company (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: Quadruple | Purpose: Treatment
Other Study IDs: ALX0171-C203
Record Dates: First submitted 2018-01-26; First posted 2018-02-01 (Actual); Results first posted 2019-07-15 (Actual); Last update posted 2019-07-30 (Actual); Status verified 2019-07

CONDITIONS: Respiratory Syncytial Virus Lower Respiratory Tract Infection
MeSH Terms: interventions — gontivimab

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- ALX-0171 1.5 mg/kg (Experimental)
  Interventions: Biological: ALX-0171 1.5 mg/kg
- Placebo (Placebo Comparator)
  Interventions: Other: Placebo

INTERVENTIONS:
Biological: ALX-0171 1.5 mg/kg — ALX-0171 1.5 mg/kg was administered via a single inhalation once daily for 3 consecutive days.
  Arms: ALX-0171 1.5 mg/kg
Other: Placebo — Placebo was administered via a single inhalation once daily for 3 consecutive days.
  Arms: Placebo

SUMMARY:
This was a randomized, double-blind, multicenter, Phase II study (NCT03418571) designed to support the selection of an optimal dose of inhaled ALX-0171 for further clinical development, taking ethnicity into consideration.

Based on the results of the Phase IIb dose-ranging study ALX0171-C201 (RESPIRE), the Sponsor decided to discontinue ALX-0171 development in infants and to early terminate the ALX0171-C203 study.

DETAILED DESCRIPTION:
Four dose levels were planned to be evaluated in four consecutive cohorts consisting of Japanese infants and young children aged 28 days to <2 years with a gestational age ≥33 weeks who were hospitalized for and diagnosed with respiratory syncytial virus (RSV) lower respiratory tract infection (LRTI):

* Dose level 1: target dose of 1.5 mg/kg
* Dose level 2: target dose of 3.0 mg/kg
* Dose level 3: target dose of 6.0 mg/kg
* Dose level 4: target dose of 9.0 mg/kg

Each cohort was planned to consist of 15 subjects enrolled and randomly assigned to receive ALX-0171 or placebo, in an allocation ratio of 4:1 (N = 12 active versus N = 3 placebo per cohort).

Due to early termination of the trial, only enrollment of Cohort 1 could be completed as planned. For Cohort 2, only 1 subject was screened but did not meet the eligibility criteria and was considered a screen failure. Therefore, data were not available for treatment groups ALX-0171 3.0 mg/kg, 6.0 mg/kg, and 9.0 mg/kg.

Of note, in line with applicable guidelines, an Independent Data Monitoring Committee (IDMC) was assigned to monitor the study. Upon completing of Cohort 1, the IDMC reviewed the available unblinded safety data and unanimously recommended to continue the study with no changes to the protocol.

ELIGIBILITY:
Main inclusion criteria:

1. Subject was a Japanese male or female infant or young child aged 28 days to <2 years with gestational age ≥33 weeks at screening.
2. Subject was of Japanese descent, i.e., born in Japan to Japanese parents and had Japanese maternal and paternal grandparents.
3. Subject weighed between ≥3.0 kg and <15.0 kg at screening.
4. Subject was otherwise healthy, but was hospitalized for and clinically diagnosed with RSV LRTI (bronchiolitis or broncho-pneumonia), i.e., showing typical clinical signs and symptoms such as tachypnea, wheezing, cough, crackles, use of accessory muscles and/or nasal flaring.
5. Subject had a positive RSV diagnostic test within 4 days of screening.
6. Subject was expected to have to stay in the hospital for at least 24 hours (according to the Investigator's judgment at screening).
7. Symptoms likely related to RSV infection (i.e., the symptoms present needed to be probably linked to the current RSV infection according to Investigator's judgment) had appeared within 4 days of screening and were not yet improving at screening and randomization.
8. Subject fulfilled at least two of the following RSV disease severity criteria at screening and randomization:

   * Inadequate oral feeding that required feeding support (i.e., nasogastric tube or i.v. line),
   * Inadequate oxygen saturation defined as:

     * Peripheral capillary oxygen saturation (SpO2) <95% on room air, or
     * Requiring oxygen supplementation to maintain adequate oxygen saturation with documented pre-supplementation value <95%
   * Signs of respiratory distress defined as:

     * Respiratory rate ≥50 breaths per minute in infants up to 12 months of age, and ≥40 breaths per minute in children above 12 months, and/ or
     * Moderate or marked respiratory muscle retractions
9. Subject had normal psychomotor development.

Others as defined in the protocol

Main exclusion criteria:

1. Subject was known to have significant comorbidities including:

   * Genetic disorders (e.g., trisomy 21, cystic fibrosis),
   * Hemodynamically significant congenital heart disease (e.g., needing corrective therapy or inotropic support),
   * Bronchopulmonary dysplasia,
   * Any hereditary or acquired metabolic (bone) diseases,
   * Hematologic or other malignancy.
2. Subject was known to be human immunodeficiency virus (HIV)-positive. If the subject was <6 months of age, known HIV-positivity of the mother was also exclusionary.
3. Subject was known to be immunocompromised.
4. Subject had or was suspected to have an active, clinically relevant concurrent infection (e.g., bacterial pneumonia, urinary tract infection). Concurrent acute otitis media was not exclusionary.
5. Subject had significant oral and/or maxillofacial malformations which would have prevented proper positioning of the face mask.
6. Subject received invasive mechanical ventilation or non-invasive respiratory support (i.e., continuous or bilevel positive airway pressure) in the 4 weeks prior to screening.
7. During the current admission, subject was initially hospitalized in an Intensive Care Unit (ICU) setting and/or received invasive mechanical ventilation or non-invasive respiratory support (i.e., continuous or bilevel positive airway pressure).
8. Subject was critically ill and/or was expected to require invasive mechanical ventilation, non-invasive respiratory support (i.e., continuous or bilevel positive airway pressure), or high-flow oxygen therapy (HFOT) at levels not enabling nebulization therapy according to the Investigator's judgment. High-flow oxygen, with a maximum flow of 2 L/kg/min, was permitted under the following conditions:

   * used as Standard of Care outside ICU setting
   * could be removed for study drug administration (Note: oxygen flow at 2 L/minute could be provided through the nebulizer)
9. Subject had received 1 or more doses of palivizumab or treatment or prophylaxis with any RSV antiviral compound (e.g., ribavirin, i.v. immunoglobulin, or any investigational drug or vaccine for RSV [including subject's mother who had been vaccinated against RSV]) at any time prior to screening.
10. Subject was required to continue or start systemic corticosteroid therapy. Subject on a maintenance therapy of inhaled corticosteroids could continue this treatment at the usual dose. Topical corticosteroids for skin disorders were permitted.
11. Subject had clinically meaningful abnormalities on a 12-lead electrocardiogram (ECG), which according to the Investigor's judgement did not allow participation of the subject in the study. A 12-lead ECG performed within 4 days of screening was acceptable. If not available, the 12-lead ECG could be performed at the time of screening.

Others as defined in the protocol

Ages: 28 Days to 2 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 15 (Actual)
Dates: Start 2018-03-01 (Actual); Primary Completion 2018-10-24 (Actual); Study Completion 2018-10-24 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Monitor, Study Director — Ablynx NV
Locations (25):
- Japan (25):
  - Investigator Site, Aoi-ku
  - Investigator Site, Asahikawa
  - Investigator Site, Fuchu-shi
  - Investigator site, Fukuyama-shi
  - Investigator Site, Funabashi
  - Investigator site, Gifu
  - Investigator Site, Isesaki
  - Investigator Site, Kawasaki
  - Investigator Site, Koga
  - Investigator Site, Kurashiki
  - Investigator Site, Kurume-shi
  - Investigator Site, Meguro-ku
  - Investigator Site, Minamiku
  - Investigator site, Nagano
  - Investigator Site, Ōmura
  - Investigator site, Saitama-shi
  - Investigator Site, Shimotsuke-shi
  - Investigator Site, Takatsuki
  - Investigator Site, Toshima-ku
  - Investigator Site, Toyohira
  - Investigator site, Ueda
  - Investigator site, Wako
  - Investigator Site, Yachiyo
  - Investigator site 1, Yokosuka
  - Investigator site 2, Yokosuka

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Sixteen subjects were screened for Cohort 1. Of these, 15 subjects were randomized. There was 1 screen failure due to consent withdrawal.
  For Cohort 2, 1 subject was screened but considered a screen failure (consent withdrawal).
  Consent was obtained from the first subject on 1 March 2018; last subject completed the final visit on 19 October 2018
Pre-assignment Details: All randomized subjects received at least 1 administration of study drug and were included in the Safety Population.
Groups:
- ALX-0171 1.5 mg/kg: Single inhalation of ALX-0171 1.5 mg/kg once daily for 3 consecutive days.
- Placebo: Single inhalation of placebo once daily for 3 consecutive days.
Period: Overall Study
Arm/Group | ALX-0171 1.5 mg/kg | Placebo
Started | 12 | 3
Completed | 11 | 3
Not Completed | 1 | 0
Not completed — Consent withdrawn by legal guardian | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | ALX-0171 1.5 mg/kg | Placebo | Total
Number analyzed (Participants) | 12 | 3 | 15
Age, Continuous [Mean (Standard Deviation); unit: months] | 7.4 (4.65) | 3.5 (3.04) | 6.6 (4.58)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 5 | 2 | 7
  Male | 7 | 1 | 8
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 12 | 3 | 15
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 0 | 0 | 0
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Safety and Tolerability of Inhaled ALX-0171 1.5 mg/kg as Measured by the Number of Subjects With at Least 1 Serious or Non-Serious Treatment-emergent Adverse Event (TEAE).
Description: Number of subjects reported with at least 1 serious or non-serious TEAEs in the ALX-0171 1.5 mg/kg treatment group and placebo treatment group.
Time Frame: From the subject's first study drug administration until completion of the subject's last visit, an average of 4 weeks
Population: Safety Population
Measure: Number; unit: participants
Arm/Group | ALX-0171 1.5 mg/kg | Placebo
Number analyzed (Participants) | 12 | 3
participants
  At least one serious TEAE | 1 | 0
  At least one non-serious TEAE | 8 | 1

2. Primary Outcome: Safety and Tolerability of Inhaled ALX-0171 1.5 mg/kg as Measured by the Number of Serious and Non-serious TEAEs.
Description: Number of serious and non-serious TEAEs reported in the ALX-0171 1.5 mg/kg treatment group and placebo treatment group.
Time Frame: From the subject's first study drug administration until completion of the subject's last visit, an average of 4 weeks
Population: Safety Population
Measure: Number; unit: TEAE
Arm/Group | ALX-0171 1.5 mg/kg | Placebo
Number analyzed (Participants) | 12 | 3
TEAE
  Serious TEAE | 2 | 0
  Non-Serious TEAE | 18 | 1

ADVERSE EVENTS:
Time Frame: From the subject's first study drug administration until the subject's study completion/discontinuation date, an average of 4 weeks.
Arm/Group | ALX-0171 1.5 mg/kg | Placebo
All-Cause Mortality (participants affected / at risk) | 0/12 | 0/3
Serious Adverse Events (participants affected / at risk) | 1/12 | 0/3
Other Adverse Events (participants affected / at risk) | 8/12 | 1/3
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | ALX-0171 1.5 mg/kg (N=12) | Placebo (N=3)
Pneumonia hemophilus (Infections and infestations) | 1 (1) | 0 (0)
Pneumonia bacterial (Infections and infestations) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | ALX-0171 1.5 mg/kg (N=12) | Placebo (N=3)
Miliaria (Skin and subcutaneous tissue disorders) | 3 (3) | 0 (0)
Dermatitis contact (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Dermatitis diaper (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Erythema (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Upper respiratory tract infection (Infections and infestations) | 2 (2) | 0 (0)
Otitis media (Infections and infestations) | 1 (1) | 0 (0)
Otitis media acute (Infections and infestations) | 1 (1) | 0 (0)
Pneumonia bacterial (Infections and infestations) | 1 (1) | 0 (0)
Diarrhoea (Gastrointestinal disorders) | 1 (1) | 0 (0)
Gastric ulcer (Gastrointestinal disorders) | 1 (1) | 0 (0)
Iron deficiency anemia (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
Middle ear effusion (Ear and labyrinth disorders) | 1 (1) | 0 (0)
Edema (General disorders) | 1 (1) | 0 (0)
Hepatic function abnormal (Hepatobiliary disorders) | 0 (0) | 1 (1)
Myoclonus (Nervous system disorders) | 1 (1) | 0 (0)
Upper respiratory tract inflammation (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)

LIMITATIONS AND CAVEATS:
Based on the results of the Phase IIb study ALX0171-C201 (RESPIRE), the Sponsor decided to discontinue ALX-0171 development in infants and to early terminate the ALX0171-C203 study. Therefore, no data are available for the higher dose groups.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Publication of any results from this study will be according to the principles of the Declaration of Helsinki, in particular point 30, and will require prior review and written agreement of the Sponsor.

DOCUMENTS (2):
  • Statistical Analysis Plan (2018-11-28): https://cdn.clinicaltrials.gov/large-docs/71/NCT03418571/SAP_000.pdf
  • Study Protocol (2017-11-13): https://cdn.clinicaltrials.gov/large-docs/71/NCT03418571/Prot_001.pdf